CLINICAL TRIAL: NCT00457847
Title: Genetics of Primary Graft Dysfunction
Brief Title: Identifying Genetic Characteristics That Increase Risk of Primary Graft Dysfunction Following Lung Transplantation
Status: Recruiting | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Columbia University (Other); Vanderbilt University (Other); Stanford University (Other); University of Alabama at Birmingham (Other); University of Michigan (Other); Johns Hopkins University (Other); Duke University (Other); University of Pittsburgh (Other); University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: 1380; R01HL081619 (NIH)
Record Dates: First submitted 2007-04-05; First posted 2007-04-09 (Estimated); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Primary Graft Dysfunction; Lung Transplantation
Keywords: PGD
MeSH Terms: conditions — Primary Graft Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Primary graft dysfunction (PGD) is a severe lung injury that can occur in the days following lung transplant surgery. The purpose of this study is to identify genetic factors that may put someone at risk for developing PGD.

DETAILED DESCRIPTION:
PGD is a severe complication that affects up to 25% of lung transplant patients following surgery. Pulmonary edema, which is an abnormal build-up of fluid in the lungs, and hypoxemia, which is low blood oxygen levels, are two common symptoms that individuals with PGD experience. Treatment for this condition is often expensive, and it is the leading cause of death following lung transplant. Many potential donors and recipients are considered unsuitable for lung transplant because of concern for the development of PGD. Therefore, the ability to accurately predict which individuals are at risk for developing PGD may allow more lung transplants to be performed. Specific characteristics in both lung donors and recipients may play an important role in determining the risk of PGD. For example, genetic variations in how the body deals with harmful chemicals called oxidants may be associated with the development of PGD. The purpose of this study is to identify the specific genetic biomarkers in donors and recipients that put individuals at risk for developing PGD following a lung transplant.

This study will enroll individuals who are undergoing lung transplantation. Blood samples will be collected from lung donors and from participants prior to surgery, immediately following surgery, and 24 hours after surgery. Study researchers will monitor participants for 72 hours following surgery for symptoms of PGD. There will be no additional study visits.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing lung transplant surgery

Exclusion Criteria:

- Individuals undergoing multi-organ transplantation except heart/lung transplants

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients going under lung transplant or heart & lung transplants
Sampling Method: Probability Sample
Enrollment: 1150 (Estimated)
Dates: Start 2007-02; Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Primary graft dysfunction | First 72 hours post lung transplantation
  ISHLT standard definition and grading system will be used

CONTACTS AND LOCATIONS:
Overall Officials: Jason D. Christie, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Diamond JM, Akimova T, Kazi A, Shah RJ, Cantu E, Feng R, Levine MH, Kawut SM, Meyer NJ, Lee JC, Hancock WW, Aplenc R, Ware LB, Palmer SM, Bhorade S, Lama VN, Weinacker A, Orens J, Wille K, Crespo M, Lederer DJ, Arcasoy S, Demissie E, Christie JD; Lung Transplant Outcomes Group. Genetic variation in the prostaglandin E2 pathway is associated with primary graft dysfunction. Am J Respir Crit Care Med. 2014 Mar 1;189(5):567-75. doi: 10.1164/rccm.201307-1283OC. PMID 24467603